CLINICAL TRIAL: NCT05413304
Title: Feasibility of Evaluating Abemaciclib Neuropharmacokinetics of Diffuse Midline Glioma Using Intratumoral Microdialysis
Brief Title: Abemaciclib Neuropharmacokinetics of Diffuse Midline Glioma Using Intratumoral Microdialysis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 220003; 22-C-0003
Record Dates: First submitted 2022-06-09; First posted 2022-06-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-27

CONDITIONS: Glioma
Keywords: Central Nervous System; Cdk4/6; Brain Cancer; Surgical Resection
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — abemaciclib; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Abemaciclib and microdialysis monitoring (Experimental): Abemaciclib orally BID for 4.5 days followed by resection or biopsy and microdialysis catheter placement with continuous monitoring for 48 hours post-operative and genomic sampling of tissue/blood; followed by abemaciclib+temozolomide maintenance therapy
  Interventions: Drug: pre-operative abemaciclib; Device: Device for Cerebral Fluid Dialysate Collection; Device: Ashion Analytics GEM ExTra; Drug: abemaciclib + temozolomide

INTERVENTIONS:
Drug: pre-operative abemaciclib — pre-operatively for 4.5 days; 200mg twice daily (9 total doses)
Device: Device for Cerebral Fluid Dialysate Collection — post-resection or post-biopsy continuous intracerebral microdialysis sampling for 48-hours to assess CNS drug entry and targeted inhibition with abemaciclib
Device: Ashion Analytics GEM ExTra — resection/biopsy genomic sampling of tumor tissue and blood to identify therapeutic targets
Drug: abemaciclib + temozolomide — abemaciclib 150mg po BID and temozolomide 200mg/m2 po daily x 5 days in 28 day cycles (temozolomide 150mg/m2 po daily x 5 days for cycle 1)

SUMMARY:
Background:

Diffuse midline gliomas are the most aggressive brain tumors of childhood and young adults. Most people with these tumors survive less than 2 years. Researchers want to see if an anticancer drug (abemaciclib) can help.

Objective:

To see if researchers can measure how much abemaciclib is in a person's brain tumor and brain fluid after they take the drug for a few days.

Eligibility:

People aged 18 to 39 with recurrent high-grade glioma or diffuse midline glioma.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Tests of heart function

Imaging scans of the brain, with a contrast agent

Screening tests will be repeated during the study. Participants will also have chest X-rays.

Participants will take abemaciclib by mouth twice a day for 4 and a half days.

Participants will undergo surgery. They will have either a tumor biopsy (a needle will be inserted to remove a small piece of tissue) or a surgical resection (part or all of the tumor will be removed). A small tube (catheter) will be placed in their brain for 48 hours to collect fluid samples. They will have a neurological exam every few hours while the tube is in place. Two days later, the tube will be removed without surgery. Participants will stay in the hospital for about 4 days for treatment.

Based on the results of abemaciclib levels in the brain, participants may keep taking abemaciclib and another drug (temozolomide) by mouth until their cancer gets worse or they have bad side effects. While taking these two drugs, participants will come back to the clinic for follow-up routinely. They will be followed by the study for life.

DETAILED DESCRIPTION:
Background

Diffuse midline gliomas are the most aggressive brain tumors of childhood and young adults, with documented 2 year survival rates of <10%. These tumors are infiltrative midline high-grade gliomas. Treatment failure is due in part to the presence of the blood-brain barrier (BBB), which limits permeability of varied agents.

Efforts to evaluate drug delivery across the BBB in midline gliomas have been restricted to post biopsy specimens. In comparison, intracerebral microdialysis sampling of cortical tissue has been shown to be a highly effective tool in determining cortical neuropharmacokinetics (brain extracellular fluid penetration, accumulation and excretion) intratumorally and peritumorally in adult brain tumor participants. Microdialysis is underutilized in the adult brain tumor setting to evaluate chemotherapy or targeted therapy permeability.

Within the US, midline gliomas are not routinely biopsied. However, in the last several years, using modern surgical techniques, biopsy at the time of diagnosis has been performed with acceptable risks (4% mortality rate), with a feasible means to molecularly characterize the tumors; in order to identify potentially druggable targets.

One of the main attributes of disease progression/proliferation in midline gliomas is associated with dysregulation of the cell cycle. CDKN2A is the primary inhibitory brake on CDK4/6 driven signaling and is commonly deleted in glioblastoma, pancreas, bladder, breast and prostate cancer. The specific CDK4/6 inhibitor, abemaciclib, has FDA approval for the treatment of metastatic breast cancer.

This is a safety and feasibility study to evaluate pharmacokinetic and pharmacodynamic effects post abemaciclib administration in recurrent high grade glioma participants (cortical and midline tumors). We propose a trial using clinical microdialysis, placed in diffuse midline glioma tissue post biopsy, as an experimental research tool, to assess CNS drug entry and targeted inhibition with abemaciclib. These studies are focused with the overall intent to inform future clinical therapies and preclinical modeling.

Objectives:

To evaluate safety and feasibility of intratumoral microdialysis placement post high grade glioma resection or midline glioma biopsy

To evaluate safety and feasibility of brain interstitial dialysate sampling in glioma participants post abemaciclib administration

To measure intratumoral vs. systemic concentrations of abemaciclib in glioma participants post abemaciclib administration

Eligibility:

Participants must have recurrent high grade glioma or diffuse midline glioma based on clinical and/or radiologic findings

Participants with cortical high grade gliomas must have previous intra-operative pathology confirming disease

Participants must be =>18 and <= 39 years of age, at time of enrollment

Ability to swallow tablets/pills

Must have adequate organ function as per laboratory testing parameters

Abemaciclib administration must be able to begin no later than 14 days after the date of radiographic diagnosis (by T2 or FLAIR imaging)

Design:

This is a safety and feasibility study to evaluate tumor pharmacokinetics (PK) and pharmacodynamics (PD) of abemaciclib in recurrent high grade glioma and midline glioma participants in need of surgical resection or biopsy, respectively.

All participants will take abemaciclib pre-operatively for 4.5 days (9 total doses of abemaciclib) at twice daily dosing.

A maximally safe surgical resection for cortical high grade glioma or stereotactic needle biopsy for midline glioma will be performed in the OR. Microdialysis insertion (based on participant safety and surgical feasibility) will be performed post-biopsy in the OR and placement will be verified by brain CT.

Continuous microdialysis sampling will be obtained over the course of the next 48 hours, with subsequent removal of the catheter at the bedside.

After discharge from NIH inpatient, PK and PD findings will assist in determination of whether the participant will continue to receive abemaciclib therapy. If intratumoral or PK brain dialysate sampling concentrations are >10nmol/L, or PD findings suggest CDK inhibition (decreased expression of Rb and/or topoII ), then restart of abemaciclib therapy along with temozolomide will be administered for maintenance therapy post resection or biopsy.

Maintenance therapy will be abemaciclib 150mg po BID x 28 days together with temozolomide 200mg/m2 po daily x 5 days in 28 day cycles (temozolomide 150mg/m2 po daily x 5 days for cycle 1). After every 3 cycles, repeat brain MRI s will be obtained to evaluate treatment response and disease progression.

If a participant starts to exhibit signs of clinical deterioration or radiographic progression, the participant will discontinue maintenance therapy, with ongoing contact for survival approximately every 6 months (+/- 14 days) until death.

Results of the PK measurements and molecular testing will be provided to the participant s home oncologist to provide for assistance with directed therapy decisions (outside of this investigational trial).

We propose to evaluate 5 participants. The accrual ceiling will be set at 17 participants to account for screen failures and inevaluable participants.

ELIGIBILITY:
* INCLUSION CRITERIA:

  * Participants must have recurrent high grade glioma or midline glioma based on clinical and/or radiologic findings
  * Participants with cortical high grade gliomas must have previous intra-operative pathology confirming disease
  * Participants must be >= 18 and <= 39 years old at the time of enrollment
  * Ability to swallow tablets/pills

Prior Therapies:

* At least 4 weeks must have elapsed since any major surgeries, with no evidence of infections. Minimally invasive biopsies (outside of the brainstem) and central line placements are not considered major surgeries
* Participants who have received prior treatment with abemaciclib or another specific CDK4/6 inhibitor are not eligible for enrollment (ex., Ribociclib, Palbociclib - list is not all inclusive)
* Participants who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade <=1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to treatment. A washout period of at least 14 days or 4 half-lives from last disease directed therapy, whichever is shorter, is required between last chemotherapy dose and treatment.
* Participants who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and treatment.
* Adequate performance scale as defined below:
* Karnofsky >=50% within 14 days prior to enrollment.
* Adequate organ function within 14 days prior to enrollment as defined below:

Hematologic Function: Participants must have an absolute neutrophil count >=1500/microliters, hemoglobin >=9 g/dL (transfusion independent, defined as not receiving blood transfusion unless related to trauma or surgeries), and platelets >=100,000/microliters (transfusion independent, defined as not receiving platelet transfusions unless related to trauma or surgeries)

Hepatic Function: Participants must have bilirubin within 1.5 x the upper limit of normal for age, with the exception of those with Gilbert syndrome, and AST/ALT within < 3 x upper limit of normal.

Renal Function: Participants must have a creatinine clearance or radioisotope GFR >60ml/min/1.73 m2 or a normal serum creatinine.

Cardiac Function: Normal ejection fraction (ECHO or cardiac MRI) >= 53% (or the institutional normal); QTC or QTcF < 450 msec.

* Willingness to avoid grapefruit or grapefruit juice during abemaciclib administration
* Informed Consent: Ability of participant or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.
* Willingness of participant or LAR to sign a written informed consent document and co-enroll in study 03-N-0164
* The effects of abemaciclib on the developing human fetus are unknown, however CDK-inhibiting agents are known to be teratogenic. Temozolomide is a cytotoxic chemotherapeutic agent which is known to be teratogenic. For these reasons, women of child-bearing potential must agree to use a highly effective method of contraception prior to study entry, for the duration of study participation, and for 3 weeks after the last dose of abemaciclib and 6 months after temozolomide. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation.

  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
  * Woman participants of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 7 days of the first dose of abemaciclib.

Highly effective contraception include intrauterine devices (IUD), hormonal (birth control pills, injections, implants), tubal ligation, or partner s vasectomy .

--Cases of pregnancy that occur during maternal exposures to abemaciclib should be reported. If a participant or spouse/partner is determined to be pregnant following abemaciclib initiation she must discontinue treatment immediately. Data on fetal outcomes and breastfeeding are to be collected for regulatory reporting and drug safety evaluation.

-Abemaciclib administration must be able to begin no later than 14 days after the date of radiographic diagnosis (by T2 or FLAIR imaging)

EXCLUSION CRITERIA:

* Participants who cannot safely undergo a biopsy due to contraindications
* Pregnant women, or women who intent to become pregnant during the study, are excluded from this study because of the teratogenic effects of abemaciclib. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is treated on study.
* Serious preexisting medical condition(s) that would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel that would preclude adequate absorption, or preexisting Crohn s disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active bleeding diatheses or renal transplant, or psychiatric illness/social situations that would limit compliance with study requirements.
* Personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Participants with HIV who have adequate CD4 counts and who have no requirement for antiviral therapy will be eligible. NOTE: Screening is not required for enrollment.
* Requires treatment with strong/moderate CYP3A inhibitors or inducers. Participants receiving any medications or substances that are inducers or strong/moderate inhibitors of CYP3A4 are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Inability to undergo MRI and/or contraindication for MRI examinations following the MRI protocol (see Study Procedure Manual). Prosthesis or orthopedic or dental braces that would interfere with MRI.
* Refractory nausea and vomiting that would limit drug administration in the opinion of the Principal Investigator
* Known severe hypersensitivity to abemaciclib, temozolomide or any excipient of abemaciclib or temozolomide or history of allergic reactions attributed to compounds of similar chemical or biologic composition to abemaciclib and temozolomide.
* Clinical judgment by the investigator that the participant should not participate in the study

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
intra-tumoral sampling adequacy | surgery/biopsy and multiple timed retrievals 2 - 48 hours post catheter insertion
  fraction of participants who have adequate intra-tumoral sampling
concentration of abemaciclib | intratumoral: surgery/biopsy and multiple timed retrievals 2 - 48 hours post catheter insertion; blood/systemic: surgery/biopsy, multiple timed retrievals 1-72 hours post catheter insertion, and Day 5 of every other maintenance therapy cycle
  intratumoral vs. systemic concentrations of abemaciclib post abemaciclib administration.
adverse events | Study Day 1 through 30 days after the last intervention
  fraction of participants who experience any adverse event/complication, including adverse events grades and types

SECONDARY OUTCOMES:
relationship between abemaciclib PK and PD studies on subsequent treatment and participant outcome | 10 years post-enrollment
  Descriptive results from abemaciclib PK and PD studies on subsequent treatment and participant outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Sadhana Jackson, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data will be shared from the time of upload to dbGaP.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Requests for all collected IPD data from clinical trials, conducted under a binding collaborative agreement between NCI/DCTD and a pharmaceutical/biotechnology company, that are not under DSMB monitoring must be in compliance with the terms of the binding collaborative agreement and must be approved by NCI/DCTD and the Pharmaceutical Collaborator (i.e., the NCI ETCTN Director in conjunction with the NCI/DCTD Regulatory Affairs Branch). @@@@@@Genomic IPD will be shared through dbGaP, per rules of the database, for purposes of genomic analysis.

REFERENCES:
- [Derived] Nduom EK, Glod J, Brown DA, Fagan M, Dalmage M, Heiss J, Steinberg SM, Peer C, Figg WD, Jackson S. Clinical protocol: Feasibility of evaluating abemaciclib neuropharmacokinetics of diffuse midline glioma using intratumoral microdialysis. PLoS One. 2023 Sep 8;18(9):e0291068. doi: 10.1371/journal.pone.0291068. eCollection 2023. PMID 37682953
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2022-C-0003.html